CLINICAL TRIAL: NCT05506683
Title: Pilot Implementation of a Nighttime Telemedicine and Medication Delivery Service to Increase Access to Pre-emergency Pediatric Care in Ghana
Brief Title: Improving Nighttime Access to Care and Treatment; Part 2- Ghana
Acronym: INACT2-G
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Ghana National Ambulance Service (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB202201648
Record Dates: First submitted 2022-08-17; First posted 2022-08-18 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2024-09

CONDITIONS: Pediatric ALL; Acute Disease
Keywords: Telemedicine; Healthcare Access; Nighttime
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Acute Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MotoMeds users (parent/chid participant pairs) (Experimental)
  Interventions: Other: MotoMeds pediatric telemedicine and medication delivery service (TMDS)

INTERVENTIONS:
Other: MotoMeds pediatric telemedicine and medication delivery service (TMDS) — The intervention is use of a pediatric TMDS. Eligible children experiencing acute illness are examined over the phone by EMTs who follow a set of clinical guidelines to triage, assess, and develop treatment plans for participants. To evaluate the TMDS and as a safety measure EMTs will also examine most participants in-person a their homes following the phone exam.

SUMMARY:
Globally, leading causes of death among children one month to 5 years old are pneumonia, diarrheal disease and malaria which are treatable early in the disease-course with low-cost medications. However, these diseases can progress to emergencies when access to care is delayed. In response, a telemedicine and medication delivery service (TMDS) was designed to improve nighttime access to pediatric care and treatment. The TMDS will be implemented in three distinct Ghanaian community to evaluate the clinical safety, operational feasibility of implementing,and scalability of the service.

DETAILED DESCRIPTION:
Globally, leading causes of death among children one month to 5 years old are pneumonia, diarrheal disease and malaria which are treatable early in the disease-course with low-cost medications. However, these diseases can progress to emergencies when access to care is delayed. In response, a telemedicine and medication delivery service (TMDS) called MotoMeds was designed to overcome barriers to seeking care. MotoMeds targets the nighttime period when barriers to accessing care are highest. The TMDS was initially deployed in Haiti and will now be evaluated for generalizability and portability in Ghana.

The study objectives are to assess clinical safety and logistical feasibility of the TMDS. The study population is children in Accra and Tamale. The workflow consists of parents/guardians calling the TMDS on their child's behalf, Emergency Medical Technicians (EMTs) referring severe cases to emergency services, EMTs performing a phone assessment for non-severe cases, and EMTs traveling to the child's household to perform an in-person exam, rapid diagnostic testing for malaria where indicated as per protocol, and to deliver protocolized medications for cases within a predefined delivery zone.

EMTs and the protocols/guidelines used are supervised by Ghanaian and US physicians.

Clinical safety and feasibility of the TMDS will be evaluated using patient and logistical metrics.

ELIGIBILITY:
Child Participant Inclusion Criteria:

* Child ≤ 10 years
* Has an acute medical problem
* Provides written assent (if 10 years and receives a household visit)

Child Participant Exclusion Criteria:

* Child > 10 years
* Child does not have an acute medical problem
* Medical problem involves physical trauma or mental health
* Refusal of written assent (if 10 years and receives a household visit)

Parent/Guardian Participant Inclusion Criteria:

* Calls MotoMeds during operating hours
* Parent/guardian of a patient participant meeting inclusion criteria
* Adult (18 years or older)
* Provides written consent (household visit) or a waiver of documentation of consent (no household visit)

Parent/Guardian Participant Exclusion Criteria:

* Age < 18 years
* No written consent or waiver of documentation of consent
* Corresponding child does not meet inclusion criteria

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1239 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
The rate of guideline adherence at the call center. | 1 day
  Establish the rates of provider adherence to the TMDS clinical guidelines while performing assessments and generating treatment plans at the call center. Points of non-adherence will include severity assessments, missed danger signs and non-indicated or missed antibiotic prescriptions.

SECONDARY OUTCOMES:
The rate of guideline adherence at the household. | 1 day
  Establish the rates of provider adherence to the TMDS clinical guidelines while performing assessments and generating treatment plans at the household. Points of non-adherence will include severity assessments, missed danger signs and non-indicated or missed antibiotic prescriptions.
Sensitivity, specificity and congruence of clinical variables | 1 day
  Determine sensitivity and specificity of each clinical variable at the call center using the in-person exam at the household as the reference standard. Establish congruence between call center and in-person assessment in terms of severity categorization, danger signs, disease type, and treatment plans.
Participant clinical status at 8-12 days | Between 8-12 days
  Determine the clinical status of participants 8-12 days following their initial contact with the TMDS. Participant families will report the status (recovered, better, same, worse, died) to TMDS staff during a follow-up phone call.

OTHER OUTCOMES:
Operational metrics: Duration of initial call and time to arrival at household | 1 hour
  Measure call duration, defined as the time elapsed from first contact between a parent/guardian and a MotoMeds call center provider until the patient's treatment plan has been relayed. Measure time to arrival at household, defined as the time elapsed from first contact between a parent/guardian and a MotoMeds call center provider until the MotoMeds team arrives at the participant's household. Data will be analyzed against benchmarks set in formative research.
Evaluate qualitative feedback from MotoMeds users | Between 8-12 days
  Parent/guardian feedback will be collected on the clinical and quality aspects of the TMDS. Both quantitative and qualitative data will be analyzed to identify strengths and weaknesses of the TMDS design.

CONTACTS AND LOCATIONS:
Overall Officials: Torben K Becker, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- National Ambulance Service, Accra, Accra Metropolitan District, Ghana

IPD SHARING:
Plan to Share IPD: Yes
The de-identified individual participant data (IDP) will be made publicly available through a data depository such as Dryad.
Time Frame: The de-identified IDP will likely be made available within 1 year of the conclusion of the study and will remain available indefinitely.
Access Criteria: The de-identified IDP will be publicly available.

REFERENCES:
- [Background] Flaherty KE, Klarman MB, Cajusma Y, Schon J, Exantus L, Beau de Rochars VM, Baril C, Becker TK, Nelson EJ. A Nighttime Telemedicine and Medication Delivery Service to Avert Pediatric Emergencies in Haiti: An Exploratory Cost-Effectiveness Analysis. Am J Trop Med Hyg. 2022 Feb 21;106(4):1063-1071. doi: 10.4269/ajtmh.21-1068. Print 2022 Apr 6. PMID 35189597
- [Background] Flaherty KE, Zakariah AN, Vescio VA, Osei-Ampofo M, Mahama MN, Agongo V, Becker TK. The state of emergency medical technician education in Ghana. Afr J Emerg Med. 2020 Sep;10(3):107-110. doi: 10.1016/j.afjem.2020.01.009. Epub 2020 Mar 7. PMID 32923318
- [Derived] Flaherty KE, Mahama MN, Klarman MB, Anane-Binfoh NA, Patel MD, Smith NJ, Osei-Ampofo M, Mathelier M, Nelson EJ, Zakariah AN, Afaa TJ, Becker TK. Applying the ADAPT guidance to implement a telemedicine and medication delivery service in a malaria-endemic setting: A prospective cohort study. Trop Med Int Health. 2025 Mar;30(3):181-192. doi: 10.1111/tmi.14081. Epub 2025 Jan 16. PMID 39815954
- See also: MotoMeds website — http://motomeds.org

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT05506683/Prot_SAP_000.pdf